CLINICAL TRIAL: NCT05418907
Title: Exendin PET/CT for Paragangliomas
Brief Title: Exendin PET/CT for Imaging of Paragangliomas
Acronym: ENTRAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-000194-93
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Paraganglioma
MeSH Terms: conditions — Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with confirmed paraganglioma: 10 patients with confirmed PGL who have undergone CT, somatostatin receptor (SSTR) PET/CT and 18F-FDG PET/CT (as standard diagnostic procedures) and are scheduled for surgery.
  Interventions: Radiation: 68Ga-NODAGA-exendin-4 PET/CT

INTERVENTIONS:
Radiation: 68Ga-NODAGA-exendin-4 PET/CT — PET/CT imaging 1 hour after injection of 100 MB 68Ga-NODAGA-exendin-4

SUMMARY:
Functional imaging of paragangliomas (PGLs) is not unequivocal. Existing functional imaging modalities show good but variable results in PGLs, warranting the search for additional molecular imaging targets. Investigators aim to evaluate the glucagon-like peptide 1 receptor (GLP-1R) as a novel target for molecular imaging of PGLs. For this purpose investigators will use the tracer 68Ga-NODAGA-exendin 4 for positron emission tomography/computed tomography (PET/CT) imaging.

DETAILED DESCRIPTION:
Rationale:

Functional imaging of paragangliomas (PGLs) is not unequivocal. Existing functional imaging modalities show good but variable results in PGLs, warranting the search for additional molecular imaging targets. Investigators aim to evaluate the glucagon-like peptide 1 receptor (GLP-1R) as a novel target for molecular imaging of PGLs. For this purpose investigators will use the tracer 68Ga-NODAGA-exendin 4 for positron emission tomography/computed tomography (PET/CT) imaging.

Objective:

The primary objective is to examine the feasibility of 68Ga-exendin-4 PET/CT for localization and functional characterization of PGLs.

Study design:

In this prospective pilot imaging study 68Ga-exendin-4 PET/CT will be performed in 10 patients with confirmed PGL who have undergone CT, somatostatin receptor (SSTR) PET/CT and 18F-FDG PET/CT (as standard diagnostic procedures) and are scheduled for surgery. 100 ± 10 MBq 68Ga-NODAGA-exendin-4 will be administered to 10 patients in total. In the first 5 patients PET/CT imaging will be performed 1, 2 and 4 hours after injection to determine the optimal imaging timepoint for the remainder of the patients, which will be applied in the remaining patients.

The images will be reconstructed and evaluated by a nuclear medicine physician who is blinded to the results of the CT, SSTR PET/CT and 18F-FDG PET/CT to assess tumor detection. Additionally, quantitative analysis of 68Ga-exendin-4, SSTR PET and 18F-FDG PET/CT images will be performed. After the patients have undergone surgery, immunohistochemical analysis of surgical specimens will be performed to assess GLP-1R expression, which will be compared with in vivo tracer uptake.

ELIGIBILITY:
Inclusion Criteria:

* Proven sympathetic PGL with a single tumor detected using standard diagnostic imaging
* No evidence of metastatic disease
* CT, SSTR PET/CT and 18F-FDG PET/CT performed (golden standard diagnostic imaging)
* Scheduled for surgery
* Able to sign informed consent

Exclusion Criteria:

* Breast feeding
* Pregnancy or the wish to become pregnant within 1 month
* Calculated creatinine clearance below 40ml/min
* Evidence of other malignancy than PGL in conventional imaging (suspicious liver, bone and lung lesions)
* Age < 18 years
* Not able to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with biochemically proven PGL
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
detection rate of PGL's using 68Ga-exendin-4 PET/CT | 1 year
  Detection based on visual inspection of PET/CT images

SECONDARY OUTCOMES:
optimal timepoint for imaging PGLs using 68Ga-exendin-4 PET/CT | After inclusion of the first 5 patients (up to 6 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided